CLINICAL TRIAL: NCT02612662
Title: A Randomized, Single-blind, Placebo-controlled Study to Assess the Safety, Tolerability and Pharmacokinetics of AZD4076 Tetracosasodium Following Single-ascending Dose Administration to Healthy Male Subjects
Brief Title: A Study to Assess the Safety and Tolerability of Single Doses of AZD4076 in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: D5590C00001
Record Dates: First submitted 2015-11-17; First posted 2015-11-24 (Estimated); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Non-alcoholic Steatohepatitis (NASH)
Keywords: AZD4076; Healthy male subjects; Safety; Subcutaneous; Tolerability
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (6):
- Cohort 1 (Experimental): Subjects will be fasted for at least 10 hours before dosing and until 4 hours after dosing of a single dose of AZD4076 tetracosasodium or placebo (high doses may be fractionated)
  Interventions: Drug: AZD4076; Drug: Placebo
- Cohort 2 (Experimental): Subjects will be fasted for at least 10 hours before dosing and until 4 hours after dosing of a single dose of AZD4076 tetracosasodium or placebo (high doses may be fractionated)
  Interventions: Drug: AZD4076; Drug: Placebo
- Cohort 3 (Experimental): Subjects will be fasted for at least 10 hours before dosing and until 4 hours after dosing of a single dose of AZD4076 tetracosasodium or placebo (high doses may be fractionated)
  Interventions: Drug: AZD4076; Drug: Placebo
- Cohort 4 (Experimental): Subjects will be fasted for at least 10 hours before dosing and until 4 hours after dosing of a single dose of AZD4076 tetracosasodium or placebo (high doses may be fractionated)
  Interventions: Drug: AZD4076; Drug: Placebo
- Cohort 5 (Experimental): Subjects will be fasted for at least 10 hours before dosing and until 4 hours after dosing of a single dose of AZD4076 tetracosasodium or placebo (high doses may be fractionated)
  Interventions: Drug: AZD4076; Drug: Placebo
- Cohort 6 (Experimental): Subjects will be fasted for at least 10 hours before dosing and until 4 hours after dosing of a single dose of AZD4076 tetracosasodium or placebo (high doses may be fractionated)
  Interventions: Drug: AZD4076; Drug: Placebo

INTERVENTIONS:
Drug: AZD4076 — Subcutaneous (SC) administration of single ascending doses; there will be no more than 2 mL per syringe/injection
Drug: Placebo — Subcutaneous (SC) administration of single ascending doses; there will be no more than 2 mL per syringe/injection

SUMMARY:
This is a first-in-human (FIH) study designed to evaluate the safety, tolerability, and pharmacokinetics (PK) of AZD4076 tetracosasodium in healthy male subjects at increasing single doses

DETAILED DESCRIPTION:
This is a Phase 1, randomized, first-in-human (FIH) study to assess the safety, tolerability, and pharmacokinetics (PK) of AZD4076 tetracosasodium following subcutaneous (SC) administration in healthy male subjects at increasing single doses

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated, written informed consent prior to any study specific procedures
2. Healthy male subjects aged 18 - 50 years with suitable veins for cannulation or repeated venipuncture
3. Have a body mass index (BMI) between 18 and 30 kg/m2 inclusive and weigh at least 50 kg and no more than 100 kg inclusive
4. Provision of signed, written and dated informed consent for optional genetic research

Exclusion Criteria:

1. History or presence of any clinically significant disease or disorder which, in the opinion of the Investigator, may either put the subject at risk because of participation in the study, or influence the results or the subject's ability to participate in the study
2. History or presence of hepatic or renal disease, or any other condition known to interfere with distribution, metabolism, or excretion of drugs
3. History or presence of significant neurological or psychiatric disease/mental illness (as judged by the investigator)
4. Suspicion of or known Gilbert's syndrome based on liver function tests
5. Any clinically significant illness, medical/surgical procedure, or trauma within 4 weeks of the administration of IMP
6. Any clinically significant abnormalities in clinical chemistry, hematology, or urinalysis results, as judged by the investigator
7. Any positive result on screening for serum hepatitis B surface antigen (HBsAg), hepatitis C antibody and human immunodeficiency virus (HIV)
8. Serum Creatinine greater than the ULN.
9. Platelet count outside the normal range.
10. AST, ALT, or GGT greater than the ULN.
11. Abnormal vital signs, after 10 minutes supine rest, defined as any of the following:

    * Systolic BP (SBP) < 90mmHg or ≥ 140 mmHg
    * Diastolic BP (DBP) < 50mmHg or ≥ 90 mmHg
    * Pulse < 45 or > 85 beats per minute (bpm)
12. Any clinically significant abnormalities in rhythm, conduction or morphology of the resting ECG and any clinically significant abnormalities in the 12-lead ECG, as considered by the investigator that may interfere with the interpretation of QTc interval changes, including abnormal ST-T-wave morphology, particularly in the protocol defined primary lead or left ventricular hypertrophy
13. Prolonged QTcF > 450 ms or shortened QTcF < 340 ms or family history of long QT syndrome
14. PR(PQ) interval shortening < 120 ms (PR > 110 ms but < 120 ms is acceptable if there is no evidence of ventricular pre-excitation)
15. PR (PQ) interval prolongation (> 240 ms) intermittent second (Wenckebach block while asleep is not exclusive) or third degree AV block, or AV dissociation
16. Persistent or intermittent complete bundle branch block (BBB), incomplete bundle branch block (IBBB), or intraventricular conduction delay (IVCD) with QRS > 110 ms. Subjects with QRS > 110 ms but < 115 ms are acceptable if there is no evidence of, for example, ventricular hypertrophy or pre-excitation
17. Known or suspected history of drug abuse, as judged by the investigator
18. Current smokers or those who have smoked or used nicotine products within the 3 months prior to screening
19. History of alcohol abuse or excessive intake of alcohol, as judged by the investigator
20. Positive screen for drugs of abuse or cotinine (nicotine) at screening or admission to the unit or positive screen for alcohol on admission to the unit prior to the administration of IMP
21. History of severe allergy/hypersensitivity or ongoing clinically significant allergy/hypersensitivity, as judged by the investigator or history of hypersensitivity to drugs with a similar chemical structure or class to AZD4076 tetracosasodium
22. Excessive intake of caffeine containing drinks or food (e.g., coffee, tea), as judged by the investigator
23. Use of drugs with enzyme inducing properties such as St John's Wort within 3 weeks prior to the administration of IMP
24. Use of any prescribed or non-prescribed medication including antacids, analgesics (other than paracetamol/acetaminophen), herbal remedies, megadose vitamins (intake of 20 to 600 times the recommended daily dose) and minerals during the two weeks prior to the administration of IMP or longer if the medication has a long half-life
25. Plasma donation within one month of screening or any blood donation/blood loss > 500 mL during the 3 months prior to screening
26. Has received another new chemical entity (defined as a compound which has not been approved for marketing) within 3 months of the administration of IMP in this study. The period of exclusion begins three months after the final dose or one month after the last visit whichever is the longest.

    Note: Subjects consented and screened, but not randomized in this study or a previous phase I study, are not excluded.
27. Vulnerable subjects, e.g., kept in detention, protected adults under guardianship, trusteeship, or committed to an institution by governmental or juridical order
28. Involvement of any Astra Zeneca, PAREXEL or study site employee or their close relatives
29. Judgment by the investigator that the subject should not participate in the study if they have any ongoing or recent (i.e., during the screening period) minor medical complaints that may interfere with the interpretation of study data or are considered unlikely to comply with study procedures, restrictions and requirements
30. Subjects who are vegans or have medical dietary restrictions
31. Subjects who cannot communicate reliably with the investigator

    In addition, any of the following is regarded as a criterion for exclusion from the genetic research:
32. Previous bone marrow transplant
33. Non-leukocyte depleted whole blood transfusion within 120 days of the date of the genetic sample collection

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2015-11-24 (Actual); Primary Completion 2017-11-04 (Actual); Study Completion 2025-10-27 (Actual)

PRIMARY OUTCOMES:
The safety and tolerability of AZD4076 by assessment of blood pressure | From screening until 16 weeks postdose, up to 5 months
  To assess the safety and tolerability of single doses of AZD4076
The safety and tolerability of AZD4076 by assessment of pulse | From screening until 16 weeks postdose, up to 5 months
  To assess the safety and tolerability of single doses of AZD4076
The safety and tolerability of AZD4076 by assessment of oral temperature | From screening until 72 hours postdose
  To assess the safety and tolerability of single doses of AZD4076
The safety and tolerability of AZD4076 by assessment of electrocardiogram readings | From screening until 16 weeks postdose, up to 5 months
  To assess the safety and tolerability of single doses of AZD4076
The safety and tolerability of AZD4076 by assessment of digital electrocardiogram readings | From predose until 72 hours postdose
  To assess the safety and tolerability of single doses of AZD4076
The safety and tolerability of AZD4076 by assessment of cardiac telemetry | On Day -1 and predose until 72 hours postdose
  To assess the safety and tolerability of single doses of AZD4076 by telemetry monitoring and paper printouts
The safety and tolerability of AZD4076 by assessment of physical examination | From screening until 16 weeks postdose, up to 5 months
  This is a composite of the general appearance, skin, cardiovascular, respiratory, abdomen, head, and neck (including ears, eyes, nose, and throat), lymph nodes, thyroid, musculoskeletal and neurological systems
The safety and tolerability of AZD4076 by assessing hematology | From screening until 16 weeks postdose, up to 5 months
  To assess the safety and tolerability of single doses of AZD4076
The safety and tolerability of AZD4076 by assessing the injection site | Postdose until 72 hours
  This includes assessment of erythema/redness, swelling, induration, pruritus and pain at injection site
The safety and tolerability of AZD4076 by assessming the number of adverse events | From screening until 16 weeks postdose, up to 5 months
  To assess the safety and tolerability of single doses of AZD4076
The safety and tolerability of AZD4076 by assessing clinical chemistry | From screening until 16 weeks postdose, up to 5 months
  To assess the safety and tolerability of single doses of AZD4076
The safety and tolerability of AZD4076 by assessing urinalysis | From screening until 16 weeks postdose, up to 5 months
  To assess the safety and tolerability of single doses of AZD4076
The safety and tolerability of AZD4076 by assessing the number of participants with adverse events | From screening until 16 weeks postdose, up to 5 months
  To assess the safety and tolerability of single doses of AZD4076

SECONDARY OUTCOMES:
Observed maximum plasma concentration, taken directly from the individual concentration-time curve [Cmax] assessed for AZD4076 from the plasma data | Predose until 16 weeks postdose
  To characterize the plasma pharmacokinetics of AZD4076
Time to reach maximum concentration, taken directly from the individual concentration-time curve [tmax] assessed for AZD4076 from the plasma data | Predose until 16 weeks postdose
  To characterize the plasma pharmacokinetics of AZD4076
Terminal elimination half-life, estimated as (ln2)/λz [t1/2λz ] assessed for AZD4076 from the plasma data | Predose until 16 weeks postdose
  To characterize the plasma pharmacokinetics of AZD4076
Area under the plasma concentration-curve from time zero to 72h after drug administration [AUC(0-72h)] assessed for AZD4076 from the plasma data | Predose until 16 weeks postdose
  To characterize the plasma pharmacokinetics of AZD4076
Area under the plasma concentration-curve from time zero to the time of last quantifiable concentration [AUC(0-last)] assessed for AZD4076 from the plasma data | Predose until 16 weeks postdose
  To characterize the plasma pharmacokinetics of AZD4076
Area under plasma concentration-time curve from time zero extrapolated to infinity [AUC] assessed for AZD4076 from the plasma data | Predose until 16 weeks postdose
  To characterize the plasma pharmacokinetics of AZD4076
Apparent total clearance, estimated as dose divided by AUC [CL/F] assessed for AZD4076 from the plasma data | Predose until 16 weeks postdose
  To characterize the plasma pharmacokinetics of AZD4076
Mean Residence Time [MRT] assessed for AZD4076 from the plasma data | Predose until 16 weeks postdose
  To characterize the plasma pharmacokinetics of AZD4076
Apparent volume of distribution at terminal phase, estimated by dividing the apparent clearance (CL/F) by λz [Vz/F] assessed for AZD4076 from the plasma data | Predose until 16 weeks postdose
  To characterize the plasma pharmacokinetics of AZD4076
Dose normalized maximum plasma concentration divided by dose, calculated by dividing Cmax by the dose administered for [Cmax/D] assessed for AZD4076 from the plasma data | Predose until 16 weeks postdose
  To characterize the plasma pharmacokinetics of AZD4076
Dose normalized area under the plasma concentration-time curve from time zero to time of last quantifiable concentration, calculated by dividing AUC(0-last) by the dose administered [AUC(0 last)/D] assessed for AZD4076 from the plasma data | Predose until 16 weeks postdose
  To characterize the plasma pharmacokinetics of AZD4076
Dose normalized area under the plasma concentration-time curve from time zero extrapolated to infinity divided by dose, calculated by dividing AUC by the dose administered [AUC/D] assessed for AZD4076 from the plasma data | Predose until 16 weeks postdose
  To characterize the plasma pharmacokinetics of AZD4076
Lag-time, taken directly from the individual concentration-time curve [tlag] assessed for AZD4076 from the plasma data | Predose until 16 weeks postdose
  To characterize the plasma pharmacokinetics of AZD4076
Cumulative amount of analyte excreted in urine from time zero to the last sampling interval (72 hours) [Ae(0-t)] assessed for AZD4076 from the urine data | Predose until 72 hours postdose
  To characterize the pharmacokinetics of AZD4076 in urine
Percentage of dose excreted unchanged into the urine from time zero to the last sampling interval (72 hours), estimated by dividing Ae(0-t) by dose [fe(0-t)] assessed for AZD4076 from the urine data | Predose until 72 hours postdose
  To characterize the pharmacokinetics of AZD4076 in urine
Renal clearance, estimated by dividing Ae(0-t) by AUC(0-72) [CLR] assessed for AZD4076 from the urine data | Predose until 72 hours postdose
  To characterize the pharmacokinetics of AZD4076 in urine
Cmax assessed for AZD4076 metabolites from the plasma data | Predose until 16 weeks postdose
  To characterize the plasma pharmacokinetics of AZD4076 metabolites (longmers, shortmers, sum of longmers and shortmers and sum of AZD4076, longmers and shortmers)
tmax assessed for AZD4076 metabolites from the plasma data | Predose until 16 weeks postdose
  To characterize the plasma pharmacokinetics of AZD4076 metabolites (longmers, shortmers, sum of longmers and shortmers and sum of AZD4076, longmers and shortmers)
t1/2λz assessed for AZD4076 metabolites from the plasma data | Predose until 16 weeks postdose
  To characterize the plasma pharmacokinetics of AZD4076 metabolites (longmers, shortmers, sum of longmers and shortmers and sum of AZD4076, longmers and shortmers)
AUC(0-last) assessed forAZD4076 metabolites from the plasma data | Predose until 16 weeks postdose
  To characterize the plasma pharmacokinetics of AZD4076 metabolites (longmers, shortmers, sum of longmers and shortmers and sum of AZD4076, longmers and shortmers)
AUC(0-72h) assessed for AZD4076 metabolites from the plasma data | Predose until 16 weeks postdose
  To characterize the plasma pharmacokinetics of AZD4076 metabolites (longmers, shortmers, sum of longmers and shortmers and sum of AZD4076, longmers and shortmers)
MRT assessed for AZD4076 metabolites from the plasma data | Predose until 16 weeks postdose
  To characterize the plasma pharmacokinetics of AZD4076 metabolites (longmers, shortmers, sum of longmers and shortmers and sum of AZD4076, longmers and shortmers)
tlag assessed for AZD4076 metabolites from the plasma data | Predose until 16 weeks postdose
  To characterize the plasma pharmacokinetics of AZD4076 metabolites (longmers, shortmers, sum of longmers and shortmers and sum of AZD4076, longmers and shortmers)
Vz/F assessed for AZD4076 metabolites from the plasma data | Predose until 16 weeks postdose
  To characterize the plasma pharmacokinetics of AZD4076 metabolites (longmers, shortmers, sum of longmers and shortmers and sum of AZD4076, longmers and shortmers)
Cmax/D assessed for AZD4076 metabolites from the plasma data | Predose until 16 weeks postdose
  To characterize the plasma pharmacokinetics of AZD4076 metabolites (longmers, shortmers, sum of longmers and shortmers and sum of AZD4076, longmers and shortmers)
[AUC(0-last)/D assessed for AZD4076 metabolites from the plasma data | Predose until 16 weeks postdose
  To characterize the plasma pharmacokinetics of AZD4076 metabolites (longmers, shortmers, sum of longmers and shortmers and sum of AZD4076, longmers and shortmers)
AUC/D assessed for AZD4076 metabolites from the plasma data | Predose until 16 weeks postdose
  To characterize the plasma pharmacokinetics of AZD4076 metabolites (longmers, shortmers, sum of longmers and shortmers and sum of AZD4076, longmers and shortmers)
Ae(0-t) assessed for AZD4076 metabolites from the urine data | Predose until 72 hours postdose
  To characterize the pharmacokinetics of AZD4076 metabolites (longmers, shortmers, sum of longmers and shortmers and sum of AZD4076, longmers and shortmers)
fe(0-t) assessed for AZD4076 metabolites from the urine data | Predose until 72 hours postdose
  To characterize the pharmacokinetics of AZD4076 metabolites (longmers, shortmers, sum of longmers and shortmers and sum of AZD4076, longmers and shortmers)
CLR assessed for AZD4076 metabolites from the urine data | Predose until 72 hours postdose
  To characterize the pharmacokinetics of AZD4076 metabolites (longmers, shortmers, sum of longmers and shortmers and sum of AZD4076, longmers and shortmers)
AUC assessed for AZD4076 metabolites from the plasma data | Predose until 16 weeks postdose
  To characterize the plasma pharmacokinetics of AZD4076 metabolites (longmers, shortmers, sum of longmers and shortmers and sum of AZD4076, longmers and shortmers)
CL/F assessed for AZD4076 metabolites from the plasma data | Predose until 16 weeks postdose
  To characterize the plasma pharmacokinetics of AZD4076 metabolites (longmers, shortmers, sum of longmers and shortmers and sum of AZD4076, longmers and shortmers)

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Goldwater, MDCM, M.Sc, CPI, Principal Investigator — PAREXEL Early Phase Clinical Unit Baltimore
Locations (1):
- Research Site, Brooklyn, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal.
  All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool. Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home